CLINICAL TRIAL: NCT00128310
Title: Randomized Phase III Trial Comparing Vinorelbine vs. Gemcitabine Plus Vinorelbine in Patients With Advanced Breast Cancer, Previously Treated With Anthracyclines and Taxanes
Brief Title: Vinorelbine Versus Gemcitabine Plus Vinorelbine in Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM 2000-04
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Neoplasm Metastasis
Keywords: Drug-resistant metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Vinorelbine; Gemcitabine

ARMS (2):
- Arm A: Vinorelbine (Active Comparator): Arm A: Vinorelbine 30 mg/m2 will be administered as an intravenous infusion over 6-10 minutes on Study Days 1 and 8.
  Interventions: Drug: Vinorelbine
- Arm B: Vinorelbine and Gemcitabine (Experimental): Arm B: Vinorelbine 30 mg/m2 will be administered as an intravenous infusion over 6-10 minutes on Study Days 1 and 8. Gemcitabine will be administered following vinorelbine at a dose of 1200 mg/m2 as an intravenous infusion over 30 minutes.
  Interventions: Drug: Vinorelbine; Drug: Gemcitabine

INTERVENTIONS:
Drug: Vinorelbine
  Other Names: Navelbine
Drug: Gemcitabine
  Other Names: Gemzar
  Arms: Arm B: Vinorelbine and Gemcitabine

SUMMARY:
This is a multicenter, randomized, prospective, Phase III study in which patients with advanced breast carcinoma previously treated with anthracyclines and taxanes will be randomly assigned to receive one of two treatment options: vinorelbine (Arm A) or gemcitabine plus vinorelbine (Arm B).

DETAILED DESCRIPTION:
The investigators assume that progression-free survival mean time for patients treated with vinorelbine will be 3 months, and for patients treated with gemcitabine plus vinorelbine will be 5 months. That implies a reduction in risk ratio of 40% (Hazard ratio = 1,67). Assuming a bilateral alpha error of 0.05 and beta error of 10%, and the number of events needed if 60% of patients have progressed after 1 year, the number of patients needed per treatment arm is 114. Considering a 10% post-randomization drop-out, the final number of patients is 252 (126 per arm).

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnoses of breast cancer, with metastases.
* Metastatic lesions should not be curable with surgery or radiotherapy.
* Women of age > 18.
* To have received a previous treatment with anthracyclines and taxanes.
* A maximum of 2 previous chemotherapy treatment lines for metastatic disease.
* Previous radiotherapy is allowed, whenever the radiated area is not the only disease location.
* At least 4 weeks since the last previous antineoplastic treatment; patient must have recovered from all previous toxicities.
* Performance status < 2 in World Health Organization (WHO) scale.
* Clinically measurable, non measurable or really non measurable disease, as per Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Life expectancy of at least 12 weeks.
* Patients able to comply and to receive an adequate follow-up.
* Adequate bone marrow function: neutrophils ≥ 2 x 10^9/L; platelets ≥ 100 x 10^9/L; hemoglobin ≥ 100 g/L.
* Calcium within normal limits.
* Premenopausal women must adopt an adequate contraceptive method during the study and up to 3 months after treatment finalization.

Exclusion Criteria:

* Active infection or serious concomitant disease (investigator's criteria).
* Clinical evidence of metastases in the central nervous system (CNS).
* Blastic bone lesions as only disease.
* Previous neurological toxicity grade 3-4 National Cancer Institute (NCI) Common Toxicity Criteria (CTC) v.2.0.
* Previous treatment with gemcitabine and/or vinorelbine.
* More than 2 previous chemotherapy treatment lines for metastatic disease.
* Abnormal liver function (bilirubin > 2.0-fold upper normal limit (UNL); alanine transaminase (ALT) and aspartate transaminase (AST) >2.5-fold UNL). In patients with hepatic metastasis, a value of ALT and AST of up to 5-fold UNL is permitted.
* Unpaired renal function (creatinine > 2.0 mg/dL).
* Pregnancy or lactating.
* Treatment with any investigational agent in the previous 4 weeks.
* Second malignancy (except for cervix carcinoma in situ or skin carcinoma - no melanoma- with an adequate treatment). Previous malignancies are allowed if disease-free survival is superior to 5 years, except for renal carcinoma or melanoma.
* Males.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2001-01-18 (Actual); Primary Completion 2006-08-15 (Actual); Study Completion 2008-01-24 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Through study completion, an average of 1 year
  Progression-free survival is calculated as the time from randomization to the first observation of disease progression or date of death (whichever occurs earlier). Progression-free survival time will be censored at the time of the most recent information for patients who are still alive at the time of the last visit.

SECONDARY OUTCOMES:
The Number of Participants Who Experienced Adverse Events (AE) | Through study completion, an average of 1 year
  Safety was assessed by standard clinical and laboratory tests. Adverse events grade were defined by the NCI CTCAE v2.0.
Objective Response Rate (ORR) | Through study completion, an average of 1 year
  Tumor response will be assessed using RECIST criteria. The best response across all treatment will be recorded. ORR is defined as the percentage of patients with a complete or partial response out of the patients who had measurable disease at baseline.
Response Duration (RD) | Through study completion, an average of 1 year
  RD is defined as the time from the date when the measurement criteria are met for complete response (CR) or partial response (PR) (whichever status is recorded first) until the date of first observation of disease progression or death occurred. For responding patients not known to have died as of the data cut-off date and who do not have progression, duration of response will be censored at the date of last visit with adequate assessment. For responding patients who receive subsequent anticancer therapy (after discontinuation from the study treatment) prior to progression, duration of response will be censored at the date of last visit with adequate assessment prior to the initiation of post-discontinuation anticancer therapy.
Overall Survival (OS) | Through study completion, an average of 1 year
  OS was defined as the time elapsed from first treatment until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital San Carlos, Madrid
Locations (2):
- Spanish Breast Cancer Research Group (GEICAM), San Sebastián de los Reyes, Madrid, Spain
- Grupo Andino de Investigación en Oncología (GAICO), Valencia, Venezuela

REFERENCES:
- [Derived] Martin M, Ruiz A, Munoz M, Balil A, Garcia-Mata J, Calvo L, Carrasco E, Mahillo E, Casado A, Garcia-Saenz JA, Escudero MJ, Guillem V, Jara C, Ribelles N, Salas F, Soto C, Morales-Vasquez F, Rodriguez CA, Adrover E, Mel JR; Spanish Breast Cancer Research Group (GEICAM) trial. Gemcitabine plus vinorelbine versus vinorelbine monotherapy in patients with metastatic breast cancer previously treated with anthracyclines and taxanes: final results of the phase III Spanish Breast Cancer Research Group (GEICAM) trial. Lancet Oncol. 2007 Mar;8(3):219-25. doi: 10.1016/S1470-2045(07)70041-4. PMID 17329192
- See also: Click here for more information about this study — http://www.geicam.org